CLINICAL TRIAL: NCT01367912
Title: Timing of Estrogen Support During the Luteal Phase of IVF / Intracytoplasmic Sperm Injection Cycle: a Randomized Controlled Trial
Brief Title: Timing of Estrogen Support During the Luteal Phase of in Vitro Fertilization (IVF)/Intracytoplasmic Sperm Injection (ICSI) Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Institutional review board, Zekai Tahir Burak Maternity and Teaching Hospital, Murat ÖZEL, M.D.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZTB
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2008-11

CONDITIONS: Infertility
Keywords: Luteal phase support; estradiol supplementation; IVF/ICSI; clinical pregnancy rate
MeSH Terms: conditions — Infertility | interventions — Estradiol; estradiol, estriol drug combination; Tablets

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Progesterone only group (No Intervention): received a single daily application of vaginal progesterone gel beginning from the day of OPU and continued at least until pregnancy was ruled out by a negative serum ß-hCG measurement performed on the 14th day after embryo transfer with no E2 added
- Progesterone+Early Estradiol group (Active Comparator): received 2 mg estradiol tablets orally two times daily beginning from the first day after hCG injection, in addition to vaginal progesterone gel
  Interventions: Drug: estradiol tablet
- Progesterone+Late estradiol group (Active Comparator): received 2 mg estradiol tablets orally two times daily beginning from the fifth day after hCG injection, in addition to vaginal progesterone gel
  Interventions: Drug: estradiol tablet

INTERVENTIONS:
Drug: estradiol tablet — received 2 mg estradiol tablets orally two times daily beginning from the first day after hCG injection, in addition to vaginal progesterone gel
  Other Names: estrofem 2 mg tablet, Novo Nordisk, Bagsvaerd, Denmark
  Arms: Progesterone+Early Estradiol group
Drug: estradiol tablet — received 2 mg estradiol tablets orally two times daily beginning from the fifth day after hCG injection, in addition to vaginal progesterone gel.
  Other Names: estrofem 2 mg tablet, Novo Nordisk, Bagsvaerd, Denmark
  Arms: Progesterone+Late estradiol group

SUMMARY:
To test the hypothesis that adding estradiol (E2) to progesterone supplementation later in the luteal phase of in vitro fertilization (IVF)/intracytoplasmic sperm injection (ICSI) cycles, rather than earlier in the luteal phase, improves clinical pregnancy rates (PRs).

DETAILED DESCRIPTION:
Several studies reported that elevated E2 may have a detrimental effect on endometrial receptivity and embryo. This conflict was the starting point of our study. The investigators thought that this luteal decrease in E2 level could be prevented by adding estradiol just before the receptivity window is open, instead of adding earlier in the luteal phase which could result in defective embryo implantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients on long GnRH agonist protocol with controlled ovarian hyperstimulation who were seen in our IVF clinic between February and November 2008, and who have E2 levels on the day of hCG administration >2500 pg/dl

Exclusion Criteria:

* Presence of azoospermia requiring testicular sperm extraction procedure
* endometriosis greater than stage II
* unilateral oophorectomy, polycystic ovarian syndrome (PCOS)
* secondary infertility
* age greater than 40 yrs and a basal follicle stimulating hormone (FSH) level higher than 12 mIU/ml were exclusion criteria

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 301 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | sixth gestational week.
  Clinical pregnancies were detected with the confirmation of positive fetal cardiac activities by transvaginal sonography in the sixth gestational week.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Mollamahmutoğlu, MD, Study Director — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity and Teaching Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Ubaldi F, Bourgain C, Tournaye H, Smitz J, Van Steirteghem A, Devroey P. Endometrial evaluation by aspiration biopsy on the day of oocyte retrieval in the embryo transfer cycles in patients with serum progesterone rise during the follicular phase. Fertil Steril. 1997 Mar;67(3):521-6. doi: 10.1016/s0015-0282(97)80080-5. PMID 9091341
- [Background] Kolibianakis EM, Devroey P. The luteal phase after ovarian stimulation. Reprod Biomed Online. 2002;5 Suppl 1:26-35. doi: 10.1016/s1472-6483(11)60214-9. PMID 12537779
- [Background] Fauser BC, Devroey P. Reproductive biology and IVF: ovarian stimulation and luteal phase consequences. Trends Endocrinol Metab. 2003 Jul;14(5):236-42. doi: 10.1016/s1043-2760(03)00075-4. PMID 12826330
- [Background] Devreker F, Govaerts I, Bertrand E, Van den Bergh M, Gervy C, Englert Y. The long-acting gonadotropin-releasing hormone analogues impaired the implantation rate. Fertil Steril. 1996 Jan;65(1):122-6. PMID 8557126
- [Background] Daya S, Gunby J. Luteal phase support in assisted reproduction cycles. Cochrane Database Syst Rev. 2004;(3):CD004830. doi: 10.1002/14651858.CD004830. PMID 15266541
- [Background] Pritts EA, Atwood AK. Luteal phase support in infertility treatment: a meta-analysis of the randomized trials. Hum Reprod. 2002 Sep;17(9):2287-99. doi: 10.1093/humrep/17.9.2287. PMID 12202415
- [Background] Jee BC, Suh CS, Kim SH, Kim YB, Moon SY. Effects of estradiol supplementation during the luteal phase of in vitro fertilization cycles: a meta-analysis. Fertil Steril. 2010 Feb;93(2):428-36. doi: 10.1016/j.fertnstert.2009.02.033. Epub 2009 Apr 1. PMID 19342034
- [Background] Gelbaya TA, Kyrgiou M, Tsoumpou I, Nardo LG. The use of estradiol for luteal phase support in in vitro fertilization/intracytoplasmic sperm injection cycles: a systematic review and meta-analysis. Fertil Steril. 2008 Dec;90(6):2116-25. doi: 10.1016/j.fertnstert.2007.10.053. Epub 2008 Jan 7. PMID 18178194
- [Background] Kolibianakis EM, Venetis CA, Papanikolaou EG, Diedrich K, Tarlatzis BC, Griesinger G. Estrogen addition to progesterone for luteal phase support in cycles stimulated with GnRH analogues and gonadotrophins for IVF: a systematic review and meta-analysis. Hum Reprod. 2008 Jun;23(6):1346-54. doi: 10.1093/humrep/den115. Epub 2008 Apr 11. PMID 18408017
- [Background] Buvat J, Marcolin G, Guittard C, Dehaene JL, Herbaut JC, Louvet AL. [Luteal support after administration of an LHRH analog for in vitro fertilization. Superiority of vaginal progesterone in comparison with oral progesterone]. Presse Med. 1990 Mar 24;19(11):527. No abstract available. French. PMID 2138757
- [Background] Farhi J, Weissman A, Steinfeld Z, Shorer M, Nahum H, Levran D. Estradiol supplementation during the luteal phase may improve the pregnancy rate in patients undergoing in vitro fertilization-embryo transfer cycles. Fertil Steril. 2000 Apr;73(4):761-6. doi: 10.1016/s0015-0282(99)00632-9. PMID 10731538
- [Background] Bergh PA, Navot D. The impact of embryonic development and endometrial maturity on the timing of implantation. Fertil Steril. 1992 Sep;58(3):537-42. doi: 10.1016/s0015-0282(16)55259-5. PMID 1521649
- [Background] Muasher S, Acosta AA, Garcia JE, Jones GS, Jones HW Jr. Luteal phase serum estradiol and progesterone in in vitro fertilization. Fertil Steril. 1984 Jun;41(6):838-43. doi: 10.1016/s0015-0282(16)47895-7. PMID 6427017
- [Background] Yang JH, Chen HF, Lien YR, Chen SU, Ho HN, Yang YS. Elevated E2: oocyte ratio in women undergoing IVF and tubal ET. Correlation with a decrease in the implantation rate. J Reprod Med. 2001 May;46(5):434-8. PMID 11396368
- [Background] Valbuena D, Martin J, de Pablo JL, Remohi J, Pellicer A, Simon C. Increasing levels of estradiol are deleterious to embryonic implantation because they directly affect the embryo. Fertil Steril. 2001 Nov;76(5):962-8. doi: 10.1016/s0015-0282(01)02018-0. PMID 11704118
- [Background] Smitz J, Bourgain C, Van Waesberghe L, Camus M, Devroey P, Van Steirteghem AC. A prospective randomized study on oestradiol valerate supplementation in addition to intravaginal micronized progesterone in buserelin and HMG induced superovulation. Hum Reprod. 1993 Jan;8(1):40-5. doi: 10.1093/oxfordjournals.humrep.a137871. PMID 8458924
- [Background] Lukaszuk K, Liss J, Lukaszuk M, Maj B. Optimization of estradiol supplementation during the luteal phase improves the pregnancy rate in women undergoing in vitro fertilization-embryo transfer cycles. Fertil Steril. 2005 May;83(5):1372-6. doi: 10.1016/j.fertnstert.2004.11.055. PMID 15866571
- [Background] Lewin A, Benshushan A, Mezker E, Yanai N, Schenker JG, Goshen R. The role of estrogen support during the luteal phase of in vitro fertilization-embryo transplant cycles: a comparative study between progesterone alone and estrogen and progesterone support. Fertil Steril. 1994 Jul;62(1):121-5. doi: 10.1016/s0015-0282(16)56826-5. PMID 8005275
- [Background] Tay PY, Lenton EA. Inhibition of progesterone secretion by oestradiol administered in the luteal phase of assisted conception cycles. Med J Malaysia. 2003 Jun;58(2):187-95. PMID 14569738
- [Background] Smitz J, Devroey P, Camus M, Deschacht J, Khan I, Staessen C, Van Waesberghe L, Wisanto A, Van Steirteghem AC. The luteal phase and early pregnancy after combined GnRH-agonist/HMG treatment for superovulation in IVF or GIFT. Hum Reprod. 1988 Jul;3(5):585-90. doi: 10.1093/oxfordjournals.humrep.a136750. PMID 3139698
- [Background] Younis JS, Ezra Y, Sherman Y, Simon A, Schenker JG, Laufer N. The effect of estradiol depletion during the luteal phase on endometrial development. Fertil Steril. 1994 Jul;62(1):103-7. doi: 10.1016/s0015-0282(16)56823-x. PMID 8005273
- [Background] Vlahos NF, Lipari CW, Bankowski B, Lai TH, King JA, Shih IeM, Fragakis K, Zhao Y. Effect of luteal-phase support on endometrial L-selectin ligand expression after recombinant follicle-stimulating hormone and ganirelix acetate for in vitro fertilization. J Clin Endocrinol Metab. 2006 Oct;91(10):4043-9. doi: 10.1210/jc.2006-0520. Epub 2006 Jul 25. PMID 16868054
- [Background] Engmann L, DiLuigi A, Schmidt D, Benadiva C, Maier D, Nulsen J. The effect of luteal phase vaginal estradiol supplementation on the success of in vitro fertilization treatment: a prospective randomized study. Fertil Steril. 2008 Mar;89(3):554-61. doi: 10.1016/j.fertnstert.2007.04.006. Epub 2007 Aug 2. PMID 17678651
- [Background] Gorkemli H, Ak D, Akyurek C, Aktan M, Duman S. Comparison of pregnancy outcomes of progesterone or progesterone + estradiol for luteal phase support in ICSI-ET cycles. Gynecol Obstet Invest. 2004;58(3):140-4. doi: 10.1159/000079115. Epub 2004 Jun 15. PMID 15205566
- [Background] Serna J, Cholquevilque JL, Cela V, Martinez-Salazar J, Requena A, Garcia-Velasco JA. Estradiol supplementation during the luteal phase of IVF-ICSI patients: a randomized, controlled trial. Fertil Steril. 2008 Dec;90(6):2190-5. doi: 10.1016/j.fertnstert.2007.10.021. Epub 2008 Jan 14. PMID 18191847
- [Result] Pouly JL, Piekrishvili R, Beaume-BrugonF, Schubert B, Janny L. Luteal phase supplementation with oestrogens doesn't improve the IVF pregnancy rate: a randomized study. Hum Reprod 2005; 20:O- 195.
- [Result] Tonguc E, Var T, Ozyer S, Citil A, Dogan M. Estradiol supplementation during the luteal phase of in vitro fertilization cycles: a prospective randomised study. Eur J Obstet Gynecol Reprod Biol. 2011 Feb;154(2):172-6. doi: 10.1016/j.ejogrb.2010.10.003. Epub 2010 Nov 9. PMID 21067858
- [Result] Causio F, Leonetti T. Luteal phase support with estrogen and progesterone in in vitro fertilization cycles using GnRHa and FSH. Gior Ital Ostet Ginecol 1997; 19: 277-82.
- [Result] Rashidi BH, Asheghan H, Jafarabadi M, Tehrani NE. The role of estrogen supplementation during the luteal phase in in vitro fertilization-embryo transfer cycles: a comparative study between progesterone and estrogen plus progesterone support. Proceedings of the 18th World Congress on Fertility and sterility; 2004 May 23-28; Montreal, Canada. Internatioanal Congress Series; 2004.p.120-123.
- [Result] Elnashar AM, Aboul-Enein GI. Endometrial receptivity. Middle East Fertil Soc J 2004; 9 (1): 10-24).